CLINICAL TRIAL: NCT03755427
Title: Immunogenicity and Safety of an Alum-adjuvanted Inactivated H7N9 Influenza Vaccine: a Randomized, Blind, Placebo-controlled, a Phase II Clinical Trial
Brief Title: A Study of An Adjuvanted Inactivated H7N9 Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016L09902/3-2
Record Dates: First submitted 2018-11-14; First posted 2018-11-28 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: H7N9 Influenza
Keywords: H7N9

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15μg H7N9 Vaccine (Experimental): Participants will be inoculated with 2 doses of 15μg hemagglutinin antigen of H7N9 vaccine at 21-day intervals.
  Interventions: Biological: 15μg H7N9 Vaccine
- Aluminum hydroxide adjuvant (Placebo Comparator): Participants will be first inoculated with one dose of seasonal influenza vaccine and followed with one dose of aluminum hydroxide adjuvant at 21-day intervals.
  Interventions: Biological: Aluminum Hydroxide Adjuvant

INTERVENTIONS:
Biological: 15μg H7N9 Vaccine — The vaccine was a inactivated, whole virion preparation of the influenza A/Shanghai/2/2013(H7N9) virus, propagated in embryonated chicken eggs，mixed with aluminum hydroxide adjuvant.
  Arms: 15μg H7N9 Vaccine
Biological: Aluminum Hydroxide Adjuvant — The seasonal influenza vaccine was a inactivated, split virion preparation of the influenza virus, propagated in embryonated chicken eggs. The aluminum hydroxide adjuvant was 0.5ml aluminum hydroxide adjuvant.
  Arms: Aluminum hydroxide adjuvant

SUMMARY:
The aim of this study is to investigate the immunogenicity and safety of the inactivated whole-virion vaccine for teenagers and adults.

The investigators will test the vaccine in participants aged above 12 years, for a randomized, blind, placebo-controlled, clinical study. The investigators designed one dosage groups: 15 μg of hemagglutinin antigen. Control group is designed to inoculate seasonal influence vaccine and aluminum hydroxide adjuvant. Participants will receive 2 doses of vaccine at 21-day intervals. Safety up to 6 months and changes in hemagglutinin inhibition (HI) titers at 21 days after each vaccination will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 12 years, healthy population
* Subjects/ (and the guardian) informed consent, voluntarily participated and signed the informed consent form, with the ability to use thermometers, scales and to fill in diary cards as required
* To comply with the requirements of clinical trial program, receive blood test before and after immunization and cooperate with follow-up

Exclusion Criteria:

* A history of influenza A (H7N9) virus infection or suspected infection Abnormal blood routine, blood biochemistry and urine routine examination indexes
* Allergy to any component in the vaccine (allergy history of any previous vaccination), especially for egg allergy
* History of asthma, history of thyroid resection, vascular nerve edema, diabetes mellitus, hypertension can not be controlled by medicine, liver and kidney diseases or malignant tumor history
* Suffered from any serious illness, such as cancer, autoimmune disease, progressive atherosclerotic disease or complications of diabetes, chronic obstructive pulmonary disease, need oxygen therapy for acute or progressive liver or kidney disease, congestive heart-failure etc.
* History of signs disease or symptoms of neurological symptoms
* Suffering from severe chronic diseases (such as Down's syndrome, diabetes, sicklemia or neurological disorders, Green's Barre syndrome)
* Acute attacks of various acute or chronic diseases in the past 7 days
* Known or suspected of respiratory disease, acute infection or chronic disease active period, HIV infection, cardiovascular disease, severe hypertension, malignant tumor during treatment, skin diseases
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition etc
* No spleen, functional absence of spleen, and splenectomy or splenectomy without any condition
* Autoimmune diseases or immunodeficiency have been treated with immunosuppressive agents in the past 6 months
* History of epilepsy, convulsions, or a family history of psychosis
* Abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities), or obvious bruising or coagulopathy
* The blood products were received within 3 months prior to the acceptance of the vaccine
* Received a live vaccine within 14 days prior to receiving the vaccine, or received a subunit or inactivated vaccine within 7 days
* Fever within 3 days prior to vaccination, axillary temperature ≥38 ℃
* Being febrile When inoculating vaccine, axillary temperature >37.0 ℃
* Women are pregnant or in the near future planned pregnancy or pregnancy test positive
* Participants in another clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Number of Subjects Reporting Solicited and Unsolicited Adverse Events (AEs) | Continuous observation for 30 days after two inoculations
  * For each group the incidence rate of subjects with solicited AE(s) with 95% confidence interval
  * For each group the incidence rate of subjects with unsolicited AE(s) with 95% confidence interval

SECONDARY OUTCOMES:
Number of participants that presented seroconversion post injection | 21 days after two inoculations
  * Seroconvertion is defined as: prevaccination Hemagglutination-inhibition test (HI) antibody titer ≤1:10 and postvaccination HI antibody titer ≥1:40, or prevaccination HI antibody titer ≥1:10 and a postvaccination increase by a factor of four or more.
  * Participants will be collected blood post first study injection, when blood samples will be taken for HI testing
Number of participants that presented seroprotection post injection | 21 days after two inoculations
  * Seroprotection is defined as postvaccination Hemagglutination-inhibition test (HI) antibody titer ≥ 1:40.
  * Participants will be collected blood post first study injection, when blood samples will be taken for HI testing
Geometric mean of Hemagglutination-inhibition titre post first study injection | 21 days after two inoculations
  * Geometric mean of Hemagglutination-inhibition test titre will be calculated for the different groups of participants post first study injection.
  * Participants will be collected blood post first study injection, when blood samples will be taken for HI testing.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Shengli, PhD, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (1):
- Suiping Center for Disease Control and Prevention, Zhumadian, Henan, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT03755427/Prot_SAP_000.pdf